CLINICAL TRIAL: NCT00120627
Title: Efficacy of Mantram Repetition on PTSD Symptoms in Veterans
Brief Title: Mantram Repetition to Manage PTSD in Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRI 04-041
Record Dates: First submitted 2005-07-12; First posted 2005-07-18 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-08

CONDITIONS: Stress Disorders, Post Traumatic
Keywords: Randomized Controlled Trial; Intervention Study; Mindfulness; Complementary Therapy; Mind-Body Relations (Metaphysics); Spiritual Therapy; Meditation; Qualitative Analysis
MeSH Terms: conditions — Combat Disorders | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Mantram + Usual Care (Experimental): Mantram Repetition Program for PTSD delivered in this study as 6-week, 90-minute per week that targeted PTSD symptoms. It was offered as an adjunct to usual care consisting of medication and case-management.
  Interventions: Behavioral: Mantram Repetition Program (MRP) plus Usual Care; Other: Usual care consisting of medication and case management
- Arm 2: Usual Care alone (Active Comparator): Usual care alone is defined as receiving 6 weeks of medication and case management, as needed by each patient. No group meetings.
  Interventions: Other: Usual care consisting of medication and case management

INTERVENTIONS:
Behavioral: Mantram Repetition Program (MRP) plus Usual Care — The MRP teaches 3 strategies to train attention and manage symptoms: Mantram Repetition, Slowing Down and One-Pointed Attention. A "mantram" is a self-selected, sacred word or phrase that is meaningful to the participant. Slowing down refers to setting priorities and doing things carefully so one is not rushed or does not make mistakes. One-pointed attention refers to concentrating on one thing at a time (similar to mindfulness). These three tools are presented to work together synergistically and cumulatively to interrupt negative thoughts and emotional states such as anger, rage, irritability and hyper-arousal. The unique focus on spiritual words is linked to what one might call inner spiritual resources. MRP was delivered in a 6-week (90 minutes/week) group setting.
  Arms: Arm 1: Mantram + Usual Care
Other: Usual care consisting of medication and case management — Usual care consisted of case management or meeting with Veterans at least once per month and monitoring medications, if prescribed.

SUMMARY:
With ongoing war in Iraq, the incidence of posttraumatic stress disorder (PTSD) in combat veterans is increasing. Creation, implementation, and testing of new and innovative interventions are needed to provide additional options for enhancing the mental health of those with PTSD. Surveys indicate that veterans are interested in complementary approaches to health care. The purpose of this study is to determine the efficacy of the Mantram Repetition Program (MRP) delivered as a brief, 6-week, complementary and portable intervention. It includes frequent, silent repetitions of a mantram (mantra), a word or phrase with spiritual associations, to manage PTSD symptoms and improve quality of life military veterans with trauma.

DETAILED DESCRIPTION:
The Mantram Repetition Program (MRP) is an innovative, portable meditation-based group intervention. In this study, the MRP was delivered in addition to usual care (defined as case management and medication) in a 6-week (90 minutes/week) group setting. The MRP was compared to usual care only.

This 4-year study employed a mixed-methods, prospective, randomized controlled trial with qualitative phone interviews at 3 months post-intervention to explore ways that the intervention was used. Outpatient Veterans (N=146) with military-related PTSD were recruited from a single VA site and randomly assigned to the experimental arm (n=71) which consisted of usual care and the mantram program versus usual care only control group (n=76).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of PTSD, military related
* Score of greater or equal to 45 on the Clinician Administered PTSD Scale
* Read and write English
* Score of > 50 on PTSD Checklist
* Has a telephone with answering machine or voice mail to receive study messages
* Has a Case Manager assigned for usual care
* Willingness to track medications, relaxation techniques and number of case manager visit

Exclusion Criteria:

* Cognitive impairment including active psychosis, untreated bipolar disorder, dementia or personality disorder that interferes with group participation
* Presence of active, serious suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2005-11; Primary Completion 2009-02 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill E Bormann, PhD RN, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

REFERENCES:
- [Background] Bormann JE. Frequent, Silent Mantram Repetition: A Jacuzzi for the Mind. Topics in Emergency Medicine. 2005 Apr 1; 27(2):163-166.
- [Background] Bormann JE, Thorp S, Wetherell JL, Golshan S. A spiritually based group intervention for combat veterans with posttraumatic stress disorder: feasibility study. J Holist Nurs. 2008 Jun;26(2):109-16. doi: 10.1177/0898010107311276. Epub 2008 Mar 20. PMID 18356284
- [Background] Bormann JE, Smith TL, Shively M, Dellefield ME, Gifford AL. Self-monitoring of a stress reduction technique using wrist-worn counters. J Healthc Qual. 2007 Jan-Feb;29(1):45-52. doi: 10.1111/j.1945-1474.2007.tb00175.x. PMID 17518033
- [Background] Bormann JE, Smith TL, Becker S, Gershwin M, Pada L, Grudzinski AH, Nurmi EA. Efficacy of frequent mantram repetition on stress, quality of life, and spiritual well-being in veterans: a pilot study. J Holist Nurs. 2005 Dec;23(4):395-414. doi: 10.1177/0898010105278929. PMID 16251489
- [Result] Bormann JE, Hurst S, Thorp SR, Glaser D. Spiritually-Based Mantram Repetition to Manage PTSD in Veterans: A Qualitative Analysis of Use and Outcomes. [Abstract]. Annals of behavioral medicine : a publication of the Society of Behavioral Medicine. 2010 Apr 1; 39(Suppl 1):216.
- [Result] Bormann JE, Liu L, Thorp SR, Lang AJ. Spiritual wellbeing mediates PTSD change in veterans with military-related PTSD. Int J Behav Med. 2012 Dec;19(4):496-502. doi: 10.1007/s12529-011-9186-1. PMID 21874605
- [Result] Bormann JE. Spiritual well-being and PTSD symptoms in veterans: A predictive model. [Abstract]. Annals of behavioral medicine : a publication of the Society of Behavioral Medicine. 2009 Dec 1; Suppl:114.
- [Result] Bormann JE, Hurst S, Kelly A. Responses to Mantram Repetition Program from Veterans with posttraumatic stress disorder: a qualitative analysis. J Rehabil Res Dev. 2013;50(6):769-84. doi: 10.1682/JRRD.2012.06.0118. PMID 24203540
- [Result] Lang AJ, Strauss JL, Bomyea J, Bormann JE, Hickman SD, Good RC, Essex M. The theoretical and empirical basis for meditation as an intervention for PTSD. Behav Modif. 2012 Nov;36(6):759-86. doi: 10.1177/0145445512441200. Epub 2012 Jun 5. PMID 22669968
- [Result] Bormann JE, Thorp SR, Wetherell JL, Golshan S, Lang AJ. Meditation-Based Mantram Intervention for Veterans with Posttraumatic Stress Disorder: A Randomized Trial. Psychological trauma : theory, research, practice and policy. 2013 Jan 1; 5(3):259-267.
- [Derived] Bormann JE, Oman D, Walter KH, Johnson BD. Mindful attention increases and mediates psychological outcomes following mantram repetition practice in veterans with posttraumatic stress disorder. Med Care. 2014 Dec;52(12 Suppl 5):S13-8. doi: 10.1097/MLR.0000000000000200. PMID 25397817

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in January 2006 and ended in December 2009. Participants were recruited from PTSD outpatient clinics and other primary care clinics in the VA system in southern California.
Pre-assignment Details: There were 4 subjects who dropped after random assignment and before entering the interventions. Two had scheduling conflicts and could not attend the groups at the time they were offered. One was too ill. The other did not have a reason.
Groups:
- Arm 1: Mantram + Usual Care: The Mantram Repetition Program teaches 3 strategies to train attention and manage symptoms: Mantram Repetition, Slowing Down and One-Pointed Attention. A "mantram" is a self-selected, sacred word or phrase that is meaningful to the participant. Slowing down refers to setting priorities and doing things carefully so one is not rushed or does not make mistakes. One-pointed attention refers to concentrating on one thing at a time (similar to mindfulness). These three tools are presented to work together synergistically and cumulatively to interrupt negative thoughts and emotional states such as anger, rage, irritability and hyper-arousal. The unique focus on spiritual words is linked to what one might call inner spiritual resources. MRP was delivered in a 6-week (90 minutes/week) group setting.
- Arm 2: Usual Care: Usual care consisting of medication and case-management.
  Usual care consisted of medication and case management: Case management consisted of provider meetings with Veterans at least once per month and monitoring medications, if prescribed.
Period: Overall Study
Arm/Group | Arm 1: Mantram + Usual Care | Arm 2: Usual Care
Started | 71 (This is the number who enrolled and was randomly assigned to receive the Mantram Repetition Program.) | 75 (This was the number that enrolled and was randomly assigned to receive the control condition.)
Began Interventions | 69 (Two people dropped due to scheduling conflict and illness.) | 73 (Two people dropped due to scheduling conflict and an unknown reason.)
Did Not Complete Post-tx Assessments | 3 (One person had a scheduling conflict and two people were incarcerated.) | 3 (Three people dropped out but no reason given.)
Completed | 66 | 70 (Three people refused the post-assessments CAPS interview only.)
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Mantram + Medication & Case Management: Mantram Repetition Program (MRP) for PTSD delivered in this study as 6-week, 90-minute per week that targeted PTSD symptoms. It was offered as an adjunct to usual care consisting of medication and case-management. The MRP includes three strategies for training attention and managing symptoms: Mantram Repetition, Slowing Down and One-Pointed Attention. A "mantram" is a self-selected, sacred word or phrase that is meaningful to the participant. Slowing down refers to setting priorities and doing things carefully so one is not rushed or does not make mistakes. One-pointed attention refers to concentrating on one thing at a time (similar to mindfulness). These three tools were presented to work together synergistically and cumulatively to interrupt negative thoughts and emotional states.
- Control Arm: Medication & Case Management Alone: Usual care consisting of medication and case-management.
  Usual care consisting of medication and case management: Case management consists of meeting with Veterans at least once per month and monitoring medications, if prescribed.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm: Mantram + Medication & Case Management | Control Arm: Medication & Case Management Alone | Total
Number analyzed (Participants) | 71 | 75 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10.31) | 58 (9.86) | 57 (10.10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 64 | 126
  >=65 years | 9 | 11 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 68 | 74 | 142
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 16 | 36
  White | 40 | 45 | 85
  More than one race | 8 | 6 | 14
  Unknown or Not Reported | 3 | 8 | 11
Region of Enrollment [Number; unit: participants]
  United States | 71 | 75 | 146

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered Posttraumatic Stress Disorder (PTSD) Scale (CAPS) From DSM-IVTR
Description: The Clinician Administered PTSD Scale (CAPS) is used to determine PTSD symptom severity and the presence or absence of a PTSD diagnosis. The total score is obtained by summing the frequency and intensity ratings for 17 items using a 5-point scale. Scores are summed and range from 0-136. The items for frequency are rated from 0="never" to 4="daily or almost everyday." The items for intensity are rated from 0="none" to 4="extreme." Higher scores indicate greater symptom severity. Total scores greater than 45 indicate the presence of a PTSD diagnosis.
  The CAPS also has 3 subscales: 1) Criterion B (re-experiencing) has 5 items that are summed and scores range from 0 to 40; 2) Criterion C (avoidance) has 7 items that are summed and scores range from 0 to 56; and 3) Criterion D (hyper-arousal) has 5 items that are summed and scores range from 0 - 40. Higher scores indicate worse symptoms.
Time Frame: Pre-treatment and post-treatment
Population: Intent to treat analysis using Expectation-Maximization (EM) algorithm in SPSS for missing data; this is a maximum-likelihood method based on group assignment, demographic variables and clinical variables.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Mantram + Medication & Case Management (Usual Care): The Mantram Repetition Program teaches 3 strategies to train attention and manage symptoms: Mantram Repetition, Slowing Down and One-Pointed Attention. A "mantram" is a self-selected, sacred word or phrase that is meaningful to the participant. Slowing down refers to setting priorities and doing things carefully so one is not rushed or does not make mistakes. One-pointed attention refers to concentrating on one thing at a time (similar to mindfulness). These three tools are presented to work together synergistically and cumulatively to interrupt negative thoughts and emotional states such as anger, rage, irritability and hyper-arousal. The unique focus on spiritual words is linked to what one might call inner spiritual resources. MRP was delivered in a 6-week (90 minutes/week) group setting.
- Arm 2: Medication & Case Management (Usual Care Alone): Usual Care defined as receiving medication management and case management, as needed.
  Usual care consisting of medication and case management: Case management consists of meeting with Veterans at least once per month and monitoring medications, if prescribed.
Arm/Group | Arm 1: Mantram + Medication & Case Management (Usual Care) | Arm 2: Medication & Case Management (Usual Care Alone)
Number analyzed (Participants) | 71 | 75
units on a scale
  Baseline CAPS Scores | 83.08 (16.17) | 82.83 (19.44)
  Post-treatment CAPS Scores | 66.16 (23.58) | 72.59 (24.97)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Medication & Case Management (Usual Care) vs Arm 2: Medication & Case Management (Usual Care Alone); 2 group (treatment vs. control) by 2 time (pre-intervention and post-intervention) one-way ANOVA; Test type: Superiority or Other; p < 0.05, ANOVA; F (1,144) = 4.12, p < .05
Statistical Analysis 2: Comparison: Arm 1: Mantram + Medication & Case Management (Usual Care) vs Arm 2: Medication & Case Management (Usual Care Alone); Test type: Superiority or Other; p < 0.05, Fisher Exact

2. Secondary Outcome: Short-Form (SF)-12v2 Health Quality of Life (Mental Health Component Score)
Description: Short-Form (SF)-12v2 measures health-related quality of life changes in mental and physical health function. The subscale SF12 Norm-Based Mental Component Summary Score rates mental health functioning. Items include "feeling calm and peaceful, having alot of energy, feeling downhearted and blue" -- all rated on a frequency scale from 1= "all of the time" to 6="none of the time." Other items ask if emotional problems such as feeling anxious or depressed interfere with (1) "accomplishing less than you like" and (2) "not doing work or activies as carefully as usual" (yes or no). Items are weighted and summed, and then converted to a 0 to 100 scale with higher scores indicating greater improvements.
Time Frame: Pre-treatment and post-treatment
Population: Intent to treat analysis using Expectation-Maximization (EM) algorithm in SPSS to replace missing values; a maximum-likelihood method based on group assignment, demographic variables and clinical variables.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Mantram + Medication & Case Management (Usual Care): The MRP teaches 3 strategies to train attention and manage symptoms: Mantram Repetition, Slowing Down and One-Pointed Attention. A "mantram" is a self-selected, sacred word or phrase that is meaningful to the participant. Slowing down refers to setting priorities and doing things carefully so one is not rushed or does not make mistakes. One-pointed attention refers to concentrating on one thing at a time (similar to mindfulness). These three tools are presented to work together synergistically and cumulatively to interrupt negative thoughts and emotional states such as anger, rage, irritability and hyper-arousal. The unique focus on spiritual words is linked to what one might call inner spiritual resources. MRP was delivered in a 6-week (90 minutes/week) group setting.
- Arm 2: Medication & Case Management (Usual Care) Alone: Usual Care defined as receiving medication management and case management, as needed.
  Usual care consisting of medication and case management: Case management consists of meeting with Veterans at least once per month and monitoring medications, if prescribed.
Arm/Group | Arm 1: Mantram + Medication & Case Management (Usual Care) | Arm 2: Medication & Case Management (Usual Care) Alone
Number analyzed (Participants) | 71 | 75
units on a scale
  Pre-treatment Mental Health Scores | 33.15 (9.08) | 32.89 (7.85)
  Post-treatment Mental Health Scores | 36.30 (8.94) | 33.17 (7.58)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Medication & Case Management (Usual Care) vs Arm 2: Medication & Case Management (Usual Care) Alone; Intent to treat analysis using Expectation-Maximization (EM) algorithm in SPSS, a maximum-likelihood method based on group assignment, demographic variables and clinical variables; Test type: Superiority or Other; p < 0.05, ANOVA

3. Secondary Outcome: Spiritual Well-being [Functional Assessment of Chronic Illness Therapy-Spiritual Wellbeing (FACIT-Sp)]
Description: FACIT-SP a measure of existential spiritual well-being. It contains 12 items that assess levels of "feeling peaceful," "having meaning and purpose in life" and "finding comfort in faith or spiritual beliefs." Items are rated on a 5-point Likert scale: 0 = "not at all" and 4 = "very much". Scores can range from 0 to 48. Higher scores reflect greater levels of spiritual well-being.
Time Frame: Pre- & Post-Intervention
Population: Intent to treat analysis using Expectation-Maximization (EM) algorithm in SPSS, a maximum-likelihood method based on group assignment, demographic variables and clinical variables.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Mantram + Medication & Case Management (Usual Care) | Arm 2: Medication & Case Management (Usual Care) Alone
Number analyzed (Participants) | 71 | 75
units on a scale
  Baseline Spiritual Wellbeing Score | 22.30 (8.36) | 20.59 (8.27)
  Post-intervention Spiritual Wellbeing Score | 26.72 (9.04) | 20.04 (8.84)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Medication & Case Management (Usual Care) vs Arm 2: Medication & Case Management (Usual Care) Alone; 2 group (treatment vs control) by 2 time points (pre-intervention and post-intervention); Test type: Superiority or Other; p < 0.0001, ANOVA

4. Secondary Outcome: Mindfulness Attention Awareness Scale (MAAS)
Description: The Mindfulness Attention Awareness Scale (MAAS) is a 15-item questionnaire scored from 1 (almost always) to 6 (almost never) assessing individual differences in frequency of mindful states over time. Scores range from 15 to 90. Higher scores indicate greater mindful attention awareness. Mindfulness has been linked to well-being and quality of life. This questionnaire has documented content validity using factor analysis, evidence of convergent and discriminant validity, and test-retest reliability.
Time Frame: Baseline, Post-Intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Mantram + Meds & Case Management (Usual Care): The MRP teaches 3 strategies to train attention and manage symptoms: Mantram Repetition, Slowing Down and One-Pointed Attention. A "mantram" is a self-selected, sacred word or phrase that is meaningful to the participant. Slowing down refers to setting priorities and doing things carefully so one is not rushed or does not make mistakes. One-pointed attention refers to concentrating on one thing at a time (similar to mindfulness). These three tools are presented to work together synergistically and cumulatively to interrupt negative thoughts and emotional states such as anger, rage, irritability and hyper-arousal. The unique focus on spiritual words is linked to what one might call inner spiritual resources. MRP was delivered in a 6-week (90 minutes/week) group setting.
- Arm 2: Meds & Case Management (Usual Care Alone): Usual Care defined as receiving medication management and case management, as needed.
  Usual care consisting of medication and case management: Case management consists of meeting with Veterans at least once per month and monitoring medications, if prescribed.
Arm/Group | Arm 1: Mantram + Meds & Case Management (Usual Care) | Arm 2: Meds & Case Management (Usual Care Alone)
Number analyzed (Participants) | 71 | 75
units on a scale
  Baseline Mindfulness Attention Awareness | 46.60 (13.40) | 47.80 (12.02)
  Post-Intervention Mindful Attention Awareness | 50.99 (13.74) | 46.04 (13.75)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Meds & Case Management (Usual Care) vs Arm 2: Meds & Case Management (Usual Care Alone); Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Arm 1: Mantram + Meds & Case Management (Usual Care); Test type: Superiority or Other; p < 0.001, Mediation using Sobel Test

5. Secondary Outcome: Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LES-Q) General Activities
Description: Quality of Life Enjoyment & Satisfaction Questionnaire general activities scale measures quality of life and satisfaction of 14 domains on a 1 (very poor) to 5 (very good) rating scale. Scores are summed and can range from 14 to 70 with higher scores indicating greater quality of life. Domains assessed represent physical health, mood, work/volunteer activity, household activity, social relationships, family relationships, leisure time activities, ability to function in daily life, sexual interest, economic status, living/housing situation, ability to get around physically without being unsafe, ability to do work or hobbies, and overall sense of wellbeing.
Time Frame: Pre- & Post-Intervention
Population: Intent to treat analysis using Expectation-Maximization (EM) algorithm in SPSS to replace missing data, a maximum-likelihood method based on group assignment, demographic variables and clinical variables.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Mantram + Medication & Case Management (Usual Care) | Arm 2: Medication & Case Management (Usual Care) Alone
Number analyzed (Participants) | 71 | 75
units on a scale
  Baseline Quality of Life Enjoyment & Satisfaction | 35.52 (9.28) | 34.98 (9.22)
  Post-intervention Quality of Life Enjoyment & Sati | 39.34 (9.33) | 35.75 (8.45)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Medication & Case Management (Usual Care) vs Arm 2: Medication & Case Management (Usual Care) Alone; Test type: Superiority or Other; p < 0.01, ANOVA

6. Primary Outcome: PTST Checklist (PCL) Civilian Version
Description: The PTSD Checklist-Civilian is a 17 item self-report measure using a 5-point Likert scale to indicate how much one is bothered by the symptoms of PTSD from trauma. Items are rated from 0="not at all" to 5="extremely". Higher scores indicate greater severity and scores range from 17-85.
Time Frame: Pre-treatment and Post-treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Mantram + Medication & Case Management (Usual Care) | Arm 2: Medication & Case Management (Usual Care) Alone
Number analyzed (Participants) | 71 | 75
units on a scale
  Pre-treatment PCL | 61.39 (11.62) | 62.70 (10.40)
  Post-treatment PCL | 55.77 (14.30) | 60.23 (12.17)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Medication & Case Management (Usual Care) vs Arm 2: Medication & Case Management (Usual Care) Alone; 2 group (treatment vs control) by 2 time (pre-intervention and post-intervention) ANOVA; Test type: Superiority or Other; p < 0.05, ANOVA

7. Secondary Outcome: Brief Symptom Inventory 18 (BSI-18) With Subscales of Depression, Anxiety, and Somatization
Description: The Brief Symptom Inventory 18 (BSI-18) is a self-report questionnaire with three subscales representing depressive symptoms, anxiety, and somatization. Each subscale consists of 6-items rated from 0=no symptoms to 4=great deal of symptoms. Scores for each subscale are summed and each subscale ranges from 0-24 with higher scores meaning worse symptoms.
Time Frame: Pre-treatment and Post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 2: Usual Care Alone: Usual care is defined as receiving 6 weeks of medication and case management, as needed by each patient. No group meetings.
  Usual care consisting of medication and case management: Case management consists of meeting with Veterans at least once per month and monitoring medications, if prescribed.
Arm/Group | Arm 1: Mantram + Usual Care | Arm 2: Usual Care Alone
Number analyzed (Participants) | 71 | 75
units on a scale
  Pre-treatment Depression Subscale | 12.52 (5.77) | 12.32 (5.55)
  Post-treatment Depression Subscale | 10.60 (6.13) | 12.24 (6.02)
  Pre-treatment Anxiety Subscale | 12.15 (5.56) | 11.98 (5.55)
  Post-treatment Anxiety Subscale | 10.96 (5.63) | 11.51 (5.46)
  Pre-treatment Somatization Subscale | 8.74 (4.99) | 9.23 (5.40)
  Post-treatment Somatization Subscale | 7.66 (4.96) | 8.44 (5.21)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Usual Care vs Arm 2: Usual Care Alone; Depression Subscale; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Arm 1: Mantram + Usual Care vs Arm 2: Usual Care Alone; Anxiety Subscale; Test type: Superiority or Other; p = 0.31, ANOVA
Statistical Analysis 3: Comparison: Arm 1: Mantram + Usual Care vs Arm 2: Usual Care Alone; Somatization Subscale; Test type: Superiority or Other; p = 0.44, ANOVA

8. Post Hoc Outcome: Re-experiencing (Criterion B) From the Clinician Administered PTSD Scale (CAPS) Clinician Administered PTSD Scale Defined by the Diagnostic and Statistical Manual, 4th Ed, Text Revision
Description: Re-experiencing Subscale (Criterion B) assesses symptoms of persistent re-experiencing of the traumatic event. This may include recurrent, intrusive recollections of the traumatic event; recurring dreams of the event; acting or feeling as if the traumatic event were occuring; and intense psychological distress at exposure to internal or external cues that symbolize or represent the event. Items are rated by frequency on a scale of 0 (never) to 4 (daily or almost every day) and on intensity on a scale of 0 (none) to 4 (extreme, incapacitating distress). Score are summed for a total subscale score ranging from 0 to 40, higher scores indicating greater levels of symptoms.
Time Frame: Pre-treatment to Post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Mantram + Usual Care: Mantram Repetition Program (MRP) for PTSD was delivered in this study as 6-week, 90-minute per week group that targeted PTSD symptoms. It was offered as an adjunct to usual care consisting of medication and case-management.
  The MRP teaches 3 strategies to train attention and manage symptoms: Mantram Repetition, Slowing Down and One-Pointed Attention. A "mantram" is a self-selected, sacred word or phrase that is meaningful to the participant. Slowing down refers to setting priorities and doing things carefully so one is not rushed or does not make mistakes. One-pointed attention refers to concentrating on one thing at a time (similar to mindfulness). These three tools are presented to work together synergistically and cumulatively to interrupt negative thoughts and emotional states such as anger, rage, irritability and hyper-arousal. The unique focus on spiritual words is linked to what one might call inner spiritual resources.
Arm/Group | Arm 1: Mantram + Usual Care | Arm 2: Usual Care Alone
Number analyzed (Participants) | 71 | 75
units on a scale
  Pre-treatment Re-experiencing Subscale | 22.59 (6.67) | 22.47 (7.20)
  Post-treatment Re-experiencing Subscale | 16.57 (8.58) | 17.05 (8.84)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Usual Care vs Arm 2: Usual Care Alone; Post-hoc analysis; Test type: Superiority or Other; p = 0.66, ANOVA

9. Post Hoc Outcome: Avoidance (Criterion C) Subscale of the Clinician Administered PTSD Scale (CAPS) From Diagnostic and Statistical Manual, 4th Ed, Text Revision
Description: Avoidance (Criterion C) Subscale assesses symptoms of feeling detached and estranged from others; markedly diminished interest in significant activities; efforts to avoid thoughts, feelings, or conversations associated with the trauma; and efforts to avoid activities, places, or people that arouse recollections of the trauma. Items are rated by frequency on a scale of 0 (never) to 4 (daily or almost every day) and on intensity on a scale of 0 (none) to 4 (extreme, incapacitating distress). Score are summed for a total subscale score ranging from 0 to 56, higher scores indicating greater levels of symptoms.
Time Frame: Pre-treatment and Post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Mantram + Usual Care: Mantram Repetition Program for PTSD was delivered in this study as 6-week, 90-minute per week group that targeted PTSD symptoms. It was offered as an adjunct to usual care consisting of medication and case-management.
  The MRP teaches 3 strategies to train attention and manage symptoms: Mantram Repetition, Slowing Down and One-Pointed Attention. A "mantram" is a self-selected, sacred word or phrase that is meaningful to the participant. Slowing down refers to setting priorities and doing things carefully so one is not rushed or does not make mistakes. One-pointed attention refers to concentrating on one thing at a time (similar to mindfulness). These three tools are presented to work together synergistically and cumulatively to interrupt negative thoughts and emotional states such as anger, rage, irritability and hyper-arousal.
Arm/Group | Arm 1: Mantram + Usual Care | Arm 2: Usual Care Alone
Number analyzed (Participants) | 71 | 75
units on a scale
  Pre-treatment Avoidance Subscale | 32.99 (7.65) | 33.73 (9.78)
  Post-treatment Subscale | 27.25 (12.12) | 30.59 (12.83)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Usual Care; Test type: Superiority or Other; p = 0.18, ANOVA

10. Post Hoc Outcome: Hyper-arousal (Criterion D) Subscale of CAPS From Diagnostic and Statistical Manual, 4th Ed., Text Revision
Description: Hyper-arousal Subscale (Criterion D) assesses symptoms of difficulty falling or staying asleep, irritability or outbursts of anger, difficulty concentrating, hypervigilance, and exaggerated startle response. Items are rated by frequency on a scale of 0 (never) to 4 (daily or almost every day) and on intensity on a scale of 0 (none) to 4 (extreme, incapacitating distress). Scores are summed for a total subscale score ranging from 0 to 40, higher scores indicating greater levels of symptoms.
Time Frame: Pre-treatment to Post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Mantram + Usual Care | Arm 2: Usual Care Alone
Number analyzed (Participants) | 71 | 75
units on a scale
  Pre-treatment Hyperarousal Subscale | 27.56 (6.12) | 27.39 (5.56)
  Post-treatment Hyperarousal Subscale | 23.37 (7.33) | 25.27 (7.36)
Statistical Analysis 1: Comparison: Arm 1: Mantram + Usual Care vs Arm 2: Usual Care Alone; Test type: Superiority or Other; p < 0.01, ANOVA

ADVERSE EVENTS:
Time Frame: Entire study.
Groups:
- Arm 1: he MRP teaches 3 strategies to train attention and manage symptoms: Mantram Repetition, Slowing Down and One-Pointed Attention. A "mantram" is a self-selected, sacred word or phrase that is meaningful to the participant. Slowing down refers to setting priorities and doing things carefully so one is not rushed or does not make mistakes. One-pointed attention refers to concentrating on one thing at a time (similar to mindfulness). These three tools are presented to work together synergistically and cumulatively to interrupt negative thoughts and emotional states such as anger, rage, irritability and hyper-arousal. The unique focus on spiritual words is linked to what one might call inner spiritual resources. MRP was delivered in a 6-week (90 minutes/week) group setting.
- Arm 2: Usual Care defined as receiving medication management and case management, as needed.
  Usual care consisting of medication and case management: Case management consists of meeting with Veterans at least once per month and monitoring medications, if prescribed.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No